CLINICAL TRIAL: NCT00620841
Title: Gene Polymorphisms in Tacrolimus Drug Interactions in Renal Transplant Patients
Brief Title: Gene Polymorphisms in Tacrolimus Drug Interactions
Acronym: DDI-TAC
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Collaborators: Fund for Scientific Research, Flanders, Belgium (Other)
Responsible Party: Catholic University Leuven, University Hospitals, University Hospital Gasthuisberg
Other Study IDs: DDI-001
Record Dates: First submitted 2008-02-13; First posted 2008-02-22 (Estimated); Last update posted 2008-02-22 (Estimated); Status verified 2008-01

CONDITIONS: Renal Transplantation
Keywords: Tacrolimus; Renal Transplantation; genetic polymorphisms; Drug drug interactions
MeSH Terms: interventions — Genotype

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — DNA samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: Patients treated with tacrolimus and experiencing a drug interaction
  Interventions: Other: genotyping

INTERVENTIONS:
Other: genotyping — Restriction fragment lenght polymorphisms

SUMMARY:
A retrospective analysis of the influence of gene polymorphisms on drug interactions between calcineurin-inhibitors and concomitant drugs in renal transplant patients.

ELIGIBILITY:
Inclusion Criteria:

* Treatment with calcineurin-inhibitor
* Renal transplantation

Exclusion Criteria:

* Drug, alcohol addiction

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Renal transplant recipients treated with a calcineurin-inhibitor
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2007-05; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Tacrolimus exposure parameters | weeks

SECONDARY OUTCOMES:
Tacrolimus daily dosing | weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dirk R Kuypers, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Brabant, Belgium